CLINICAL TRIAL: NCT06713954
Title: Analysis of Dietary Intake in Professional Female Football Players: Variations According to Playing Position, Age, and Country
Brief Title: Analysis of Dietary Intake in Professional Female Football Players
Status: Recruiting | Type: Observational
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Blanca Roman-Viñas, MD, Professor of Health, Physical Activity and Sport, University Ramon Llull
Other Study IDs: 27-11-24
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dietary Assessment
Keywords: athlete; female; diet
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female footballers: Female footballers of varying ages, playing positions and countries
  Interventions: Behavioral: Dietary assessment

INTERVENTIONS:
Behavioral: Dietary assessment — Dietary intake data will be collected using the Snap-N-Send method, a tool with enhanced validity for assessing athlete total energy intake, where participants will take photographs of their meals and share them via WhatsApp directly with the researcher. Before the study commences, participants will receive standardised instructions on photographing food and adding details in the message such as title, portion sizes and ingredients alongside each photo to enhance data precision. The principal investigator will input these photographs with the added information into Nutritics dietary analysis software, where food weights, portion sizes, and nutritional content will be estimated and calculated. Nutritics will then calculate dependent variables and convert it into a food diary report, aggregating the three days of food diary into average intake.

SUMMARY:
This study evaluates the dietary intake of professional female footballers against nutritional guidelines, analysing differences by age, position, and location (UK vs Spain). Using a cross-sectional design, it will include 20-30 players per club from four clubs, aged 18+, collected via the Snap-N-Send method and analysed with Nutritics software. Variables include energy intake, macronutrients, and micronutrients, with data assessed using MANOVA, t-tests, and Shapiro-Wilk tests. The aim is to determine dietary adequacy and provide insights to improve nutrition education and wellbeing for female athletes.

DETAILED DESCRIPTION:
The aim of this research is to evaluate the dietary intake of female footballers against established nutritional guidelines, while analysing the variables of age, playing position and location to identify if there is a difference in intake across the groups. The study will employ an observational, descriptive, and cross-sectional research design, focusing on female footballers from professional clubs, specifically two clubs in United Kingdom and two clubs in Spain. There is an anticipated sample size of 20 to 30 participants from each club. Inclusion criteria will be female participants who are professional footballers, aged 18 and older and free of disease. Dependent variables from dietary intake will include energy intake (kcal), energy availability (kcal/kg fat free mass/day), protein (g/day), carbohydrates (g/day), fat (%), vitamin D (mg/day), calcium (mg/day) and iron (mg/day). These will be collected using the scientifically valid Snap-N-Send method and analysed with Nutritics dietary analysis software, which has been validated for assessing macronutrients and micronutrients. Independent variables will consist of age groups, playing positions, and country of origin (England or Spain). Dietary intake will be recorded through WhatsApp, with subsequent data entry and storage in Nutritics. Statistical analyses will include MANOVA, used to compare dietary data among groups, one-sample t-test to test against published recommendations and the Shapiro-Wilk test to assess normality in data distribution. This study aims to assess the adequacy of the players' dietary intake in relation to established nutritional recommendations from different backgrounds and characteristics. Furthermore, practitioners can potentially make informed decisions that improve the nutrition education given to female athletes, which contributes to their overall health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Female or assigned female at birth
* Playing football professionally
* At a sub-elite to elite standard
* Above the age of 18
* Healthy and free of disease

Exclusion Criteria:

* Active supplementation with ergogenic aids
* Active pregnancy
* No signing of the consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Age=
    * 18-24 years of age
    * 25-31 years of age
  * Playing position=
    * Defenders: Centre-backs, fullbacks, wingbacks, goalkeepers
    * Midfielders: Central midfielders, attacking midfielders, defensive midfielders
    * Wingers: Left wingers and right wingers
    * Forwards: Strikers and centre-forwards
  * Country=
    * England
    * Spain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Carbohydrates | From enrollment to the end of assessment of 3 days
  Amount of carbohydrates in grams from an average of 3 days
Energy intake | From enrollment to the end of assessment of 3 days
  Average of energy intake in calories over 3 days
Protein | From enrollment to the end of assessment of 3 days
  Average of protein in grams over 3 days
Fat | From enrollment to the end of assessment of 3 days
  Average of percentage of fat over 3 days
Energy availability | From enrollment to the end of assessment of 3 days
  Energy availability will be calculated by estimating fat-free mass (FFM) through the Boer equation, which uses weight and height. The formula for females is FFM (kg) = 0.252 × Weight (kg) + 0.473 × Height (cm) - 48.3. Total energy intake (TEI) will be determined from average daily calorie intake. Exercise energy expenditure (EEE) will be estimated based on activity duration and MET values using the Compendium of Physical Activities (Ainsworth et al., 2011). The resulting EA will be calculated using the formula: EA = (TEI - EEE) / FFM. The outcome will be an average of kcal/kg fat free mass/day over 3 days

SECONDARY OUTCOMES:
Calcium | From enrollment to the end of assessment of 3 days
  Average of calcium intake in milligrams over 3 days
Vitamin D | From enrollment to the end of assessment of 3 days
  Estimation of average of Vitamin D in micrograms over 3 days
Iron | From enrollment to the end of assessment of 3 days
  Average of iron intake in milligrams over 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Roman Viñas, PhD, Principal Investigator — Universitat Ramon Llull
Locations (1):
- Blanquerna Institute, Universitat Ramon Llull, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP